CLINICAL TRIAL: NCT02479711
Title: A Clinical Evaluation of a Glass Ionomer Cement (GIC) Based Restorative System
Brief Title: A Clinical Evaluation of a Glass Ionomer Cement (GIC) Based Restorative System Versus Bulk Filled Resin-based Composite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, elif kantar atila, Research Assisstant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dep of Pedodontics, Ege
Record Dates: First submitted 2015-04-22; First posted 2015-06-24 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Caries
Keywords: glass ionomer; bulk fill composite
MeSH Terms: interventions — Glass Ionomer Cements; EQUIA composite

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- composite restoration (Experimental): lower permanent molar with an approximal and /or occlusal carious lesion will be restored with Tetric EvoCeram Bulk Fill composite
  Interventions: Other: composite restoration
- glass ionomer cement (Active Comparator): lower permanent molar with an approximal and /or occlusal carious lesion will be restored with the glass ionomer restoration, Equia
  Interventions: Other: glass ionomer cement

INTERVENTIONS:
Other: composite restoration — The tooth will be isolated with cotton rolls and the caries will be removed. Enamel and dentin conditionings were performed with a self-etching adhesive system (Adhese One F, Ivoclar Vivadent, Liechtenstein). Bulk fill composite (Tetric EvoCeram® , Ivoclar Vivadent, Liechtenstein) will be injected in a single bulk increment of less than 4 mm to fill the preparations. The material was condensed with a flat instrument. Once set, it will be polished with finishing cups (Enhance® , Dentsply , Milford, USA). An interproximal strip will be used to finish the final contour.
  Other Names: Tetric EvoCeram Bulk fill composite
  Arms: composite restoration
Other: glass ionomer cement — The tooth will be isolated wit cotton rolls and the caries will be removed. The dentist will mix and handle the materials in accordance with the manufacturers' instructions. The material was condensed with a flat instrument. Once set, it will be polished. An interproximal strip will be used to finish the final contour. G-Coat Plus (GC, America) will be applied to the surface and margins of the restoration.
  Other Names: a high viscosity glass ionomer cement; Equia
  Arms: glass ionomer cement

SUMMARY:
The aim of the present study is to evaluate the clinical performance of EQUİA restoration material in Class II cavities comparing with a resin-based composite / dentin bonding system.

DETAILED DESCRIPTION:
35 patients at 12-year-old, who have a matched pair of permanent molars with an approximal and /or occlusal carious lesion of similar size will be included.

split -mouth design for the two restorative materials will be used. After removing the carious each patient will receive two restorations following the taking impressions to determine the cavity size.

One of the two materials will be Equia (GC Europe N.V., Leuven , Belgium), a high viscosity glass ionomer cement and the second material used will be Tetric EvoCeram Bulk Fill composite (IvoClar Vivadent), along with a dentin bonding system (AdheSe One F, Ivoclar Vivadent, Lichtenstein).

The dentist will randomly select the restorative material to be placed. The dentist will mix and handle the materials, in accordance with the manufacturers' instructions.

The clinician will use a matrix to maintain tight adaptation of the restorations.

The clinician will take impressions after the first setting reactions of the materials are done to determine the wear of the restorative materials.

Two blinded examiners who were not involved in the placement of the restorations will evaluate the restorations at six, 12 and 24 months.

Impressions will be repeated at 12 and 24 months intervals. The examiners will use the U.S Public Health Service (USPHS) Ryge criteria to evaluate the restorations.

Wear analysis will be performed with a 3 dimensional laser scanning device (Laserscan 3D, Willytec, Germany) by scanning the cast models.

The data will be analyzed using statistical software (SPSS 13.0, SPSS, Chicago). Cumulative survival rates will be estimated using the Kaplan-Meier method and long-rank-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has occlusal carious lesions in their mandibular molar teeth

Exclusion Criteria:

* Patients with extremely poor oral hygiene, severe or chronic periodontitis, or heavy bruxism habits were excluded from the study

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Wear of bulk filled resin-based composite versus high viscosity glass ionomer cement | 2 years
  using with a 3 dimensional laser scanning device by scanning cast models
Clinical performance of bulk filled resin-based composite versus high viscosity glass ionomer cement | 2 years
  in accordance with Ryge criteria

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Ersin, Study Director — Ege University; Fahinur Ertugrul, Study Chair — Ege University; Arzu Aykut- Yetkiner, Principal Investigator — Ege University; İlhan Uzel, Principal Investigator — Ege University; Elif Atila, Principal Investigator — Ege University

REFERENCES:
- [Background] Ersin NK, Candan U, Aykut A, Oncag O, Eronat C, Kose T. A clinical evaluation of resin-based composite and glass ionomer cement restorations placed in primary teeth using the ART approach: results at 24 months. J Am Dent Assoc. 2006 Nov;137(11):1529-36. doi: 10.14219/jada.archive.2006.0087. PMID 17082278
- [Background] Ryge G. Clinical criteria. Int Dent J. 1980 Dec;30(4):347-58. PMID 6935165
- [Background] Campos EA, Ardu S, Lefever D, Jasse FF, Bortolotto T, Krejci I. Marginal adaptation of class II cavities restored with bulk-fill composites. J Dent. 2014 May;42(5):575-81. doi: 10.1016/j.jdent.2014.02.007. Epub 2014 Feb 18. PMID 24561041
- [Background] Alrahlah A, Silikas N, Watts DC. Post-cure depth of cure of bulk fill dental resin-composites. Dent Mater. 2014 Feb;30(2):149-54. doi: 10.1016/j.dental.2013.10.011. Epub 2013 Nov 20. PMID 24268044
- [Background] Gurgan S, Kutuk ZB, Ergin E, Oztas SS, Cakir FY. Four-year randomized clinical trial to evaluate the clinical performance of a glass ionomer restorative system. Oper Dent. 2015 Mar-Apr;40(2):134-43. doi: 10.2341/13-239-C. Epub 2014 Oct 9. PMID 25299703